CLINICAL TRIAL: NCT06015438
Title: Physical Activity and Hidradenitis Suppurativa: A Novel Controlled Trial Investigating Functional Performance and Activity Limitations and Assessing the Benefits of an Outcome Measures Driven Exercise Program
Brief Title: Physical Activity in Hidradenitis Suppurativa (HS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Associate Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20230495
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Exercise EP Group (Experimental): Participants in this group will follow an at home personalized EP for up to 12 weeks.
  Interventions: Behavioral: Home Exercise Program
- Short EP Group (Active Comparator): Participants in this group will be enrolled in the short EP program.
  Interventions: Behavioral: Short Exercise Program

INTERVENTIONS:
Behavioral: Home Exercise Program — Participants will perform a minimum of one exercise from each of the targeted muscle groups at a frequency of every other day, for a total of 3-4 days a week of exercise with a rest day. The entire strengthening exercise routine should take approximately 25-30 minutes to perform, including rest periods. Each muscle grouping of exercises is designed to progress from minimal muscle effort required to moderate to maximal effort. Participants will use a video to perform the exercises as well as a handout with specific instructions.
  Arms: Home Exercise EP Group
Behavioral: Short Exercise Program — Participants in this group will attend one in-person visit expected to last about 60 minutes. The clinic visit will consist of standard of care procedures and tests for individuals with mild-to-severe HS .
  Arms: Short EP Group

SUMMARY:
The purpose of the study is to characterize the challenges to physical activity and exercise for HS patients and design an exercise program (EP) with evidence-based techniques and examine its outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old to 80 years old
* Have diagnosis of HS confirmed by a dermatologist
* Able to provide informed consent
* For the extended portion of the study: Classified as having moderate-to-severe HS as per the IHS-4 criteria

Exclusion Criteria:

* Individuals who are not yet adults
* Women known to be pregnant
* Prisoners
* Subjects, who in the opinion of the PI, cannot comply with the study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Strength/Endurance as Measured by 30-second chair-stand test | Baseline and up to 12 weeks
  Determines how many times a person can rise from a chair and sit down again in 30 seconds while keeping their arms crossed over their chest. The test will assess lower body strength and endurance and will be reported using a composite score of the number of times completed.
Change in Functional Strength/Endurance as measured by six-minute walk test | Baseline and up to 12 weeks
  Six-minute walk measures overall functioning capacity, and lower body muscle strength/ endurance, with a composite score reported in meters.
Change in Functional Strength as measured by hand grip strength test | Baseline and up to 12 weeks
  It is a measure of upper body muscular strength measured in kilograms.

SECONDARY OUTCOMES:
Quality of life impairment as measured by the DLQI | Baseline, up to 12 weeks
  Dermatology Life Quality Index (DLQI) has a total score ranging from 0 to 30 with the lower score indicating higher health related quality of life.
Quality of life impairment as measured by the HiSQOL | Baseline, up to 12 weeks
  Hidradenitis Suppurativa Quality of Life (HiSQOL) has a total score ranging from 0 to 68 with the lower score indicating higher health related quality of life.
Change in Physical activity as measured by the International Physical Activity Questionnaire (IPAQ) | Baseline, up to 12 weeks
  IPAQ assesses 3 types of physical activity undertaken across the 4 domains- leisure time physical activity; domestic and gardening (yard) activities; work-related physical activity; transport-related physical activity- in the previous 7 days. The 3 types of activity assessed are walking, moderate-intensity activities and vigorous-intensity activities. The result s is not reported in scales. Computation of the total score for the IPAQ requires summation of the duration (in minutes) and frequency (days) of the 3 types of activities across the 4 domains. Higher result indicates higher physical activity in the last 7 days
Change in Level of Activity as measured by the average number of steps daily | Baseline, up to 12 weeks
  Average number of steps daily will be measured with a pedometer and will be reported.
Change in Severity of HS score using the IHS-4 | Baseline, up to 12 weeks
  The International Hidradenitis Suppurativa Severity Score System (IHS4) measures HS severity as mild (0-3), moderate (4-10), severe (≥11). Higher score indicate increased severity.
Average pain as assessed by the Numerical Rating Scale (NRS) | Up to 8 weeks
  The average pain will be measured using the NRS with scores ranging from 0-10 with the higher score indicating more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No